CLINICAL TRIAL: NCT05057143
Title: The Use of Individual 3D-implants in the Reconstruction of the Chest Wall in Patients With the Tumor Lesions of the Chest Wall for the Treatment, Restoration, and Improved Quality of Life Compared to Reconstruction With Titanium Plates
Brief Title: 3D Printed Implants for the Defect Reconstruction in Patients With Chest Wall Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CWP-2021-7-3
Record Dates: First submitted 2021-09-07; First posted 2021-09-27 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Tumor of Bone; Chest Wall Tumor; Chest Wall Sarcoma; Sarcoma of Bone; Surgery; Implant Site Reaction
Keywords: Chest Wall Tumor; Surgery
MeSH Terms: conditions — Bone Neoplasms; Osteosarcoma | interventions — Bone Plates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Replacement of a defect in the chest wall with an individual implant (Experimental): A patient with a tumor lesion of the chest wall undergoes СT scan with a step width of less than 1 mm, then engineers design an individual model to replace the defect. Using a 3D printer, a model is made based on the patient's anthropometric data.
  Interventions: Device: Implants
- Replacement of a defect in the chest wall with titanium plates (Active Comparator): The use of standard titanium plates to replace the chest defect. These plates must be modeled and modified using special equipment intraoperatively, based on the characteristics of the defect after resection.
  Interventions: Device: Plates

INTERVENTIONS:
Device: Implants — 3D printed implants
  Arms: Replacement of a defect in the chest wall with an individual implant
Device: Plates — Titanium plates
  Arms: Replacement of a defect in the chest wall with titanium plates

SUMMARY:
A patient with a tumor lesion of the chest wall undergoes CT scan with a step width of less than 1 mm, then engineers design an individual model to replace the defect. Using a 3D printer, a model is made based on titanium alloy powder. Preoperative preparation takes an average of 14-21 days. The next stage is surgical treatment in the amount of resection of the chest wall with plastic defect with an individual titanium implant. In some cases, the titanium framework is separated from the pleural cavity by a polytetrafluoroethylene plate in order to seal and prevent the development of pulmonary hernias. The advantages of titanium individual prostheses include accurate matching of the implant to the size and characteristics of the defect, individual modeling allows you to repeat the anatomical features of the patient. This method helps to recreate the original shape of the chest, and most importantly, symmetrical, relatively healthy half. With the help of titanium, individualized prostheses are made based on 3D modeling, which will reduce the incidence of complications, accelerate rehabilitation and improve the quality of life of patients with tumor lesions of the chest wall. The postoperative period takes 15-30 days.

DETAILED DESCRIPTION:
A patient with a tumor lesion of the chest wall undergoes CT scan with a step width of less than 1 mm, then engineers design an individual model to replace the defect. Using a 3D printer, a model is made based on the patient's anthropometric data.

Manufacturing takes place by 3D printing on a titanium alloy powder certified for the manufacture of medical implants. The technology used is a type of SLS (Selective Laser Sintering) -technology, layer-by-layer laser melting of metal-powder compositions. The printing process begins with dividing the digital 3D model of the product into layers with a thickness of 20 to 100 microns in order to create a 2D image of each layer of the product (section). The industry standard format is STL (Stereolithography) file. This file enters a special machine software, where the information is analyzed and compared with the technical capabilities of the machine. Based on the data obtained, a production cycle of construction is launched, consisting of many cycles of building individual layers of the product.

The cycle for constructing a layer (section) consists of typical operations:

* applying a layer of powder of a given thickness to the construction plate;
* scanning by a laser beam of the section of the product layer. The laser beam is a source of heat, under the influence of which the particles of the material are sintered along the profile of the section of the model;
* lowering the platform into the depth of the construction well by an amount corresponding to the thickness of the construction layer.

The process of building products takes place in the SLM (Selective Laser Melting) chamber of the machine, filled with an inert gas argon. After construction, the product is removed from the printer chamber and sent for heat treatment, annealing, to relieve internal stresses and improve mechanical properties. After annealing, the product is separated from the platform and undergoes finishing, which combines various types of machining. The final stages of the technological process are product cleaning and technical quality control.

Preoperative preparation takes an average of 14-21 days. The next stage is surgical treatment in the amount of resection of the chest wall with plastic defect with an individual titanium implant. In all cases, the titanium framework is separated from the pleural cavity by a synthetic polyester (Dacron) plate in order to seal and prevent the development of pulmonary hernias. The advantages of titanium individual implants include accurate matching of the implant to the size and characteristics of the defect, individual modeling allows you to repeat the anatomical features of the patient. This method helps to recreate the original shape of the chest, and most importantly, symmetrical, relatively healthy half. With the help of titanium, individualized prostheses are made based on 3D modeling, which will reduce the incidence of complications, accelerate rehabilitation and improve the quality of life of patients with tumor lesions of the chest wall. The postoperative period takes 15-30 days.

ELIGIBILITY:
Inclusion Criteria:

* Malignant neoplasm of ribs, sternum and clavicle
* Malignant neoplasm of the connective and soft tissues of the chest
* Neoplasm of uncertain or unknown nature of ribs, sternum and collarbone
* Benign neoplasm of ribs, sternum and collarbone
* Tumor lesions of the chest wall of any localization, malignant and benign, as well as of an uncertain or unknown nature
* For malignant tumors: Grade 1-3
* Lack of distant metastases
* Signed informed consent

Exclusion Criteria:

* Children, women during pregnancy, childbirth, women during breastfeeding.
* Military personnel, with the exception of contract military personnel.
* Persons with mental disorders.
* Persons detained, taken into custody, serving a sentence in the form of restriction of freedom, arrest, imprisonment or administrative arrest.
* Patients with distant metastases (except for a solitary focus in the chest wall without other manifestations of the disease)
* Inoperable tumor
* The presence of another malignant tumor at the time of examination
* ECOG 4
* Having an active or chronic fungal / bacterial / viral infection
* Uncontrolled chronic diseases of the liver, kidneys in the acute stage
* Presence of metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 24 months
  Time after treatment during which no sign of cancer is found

SECONDARY OUTCOMES:
Comparison of hospitalization rate | 30 days
  Time after surgery till the end of hospitalization
Comparison of safety assessment | 24 months
  Adverse Event Assessment and Serious Adverse Event Assessment according to CTCAE 5.0
Comparison of performance status according Karnofsky scale | 24 months
  Improvement on the Karnofsky scale by 10-30 points
Comparison of pain relief according Visual Analogue Scale | 24 months
  Improvement on the Visual Analogue Scale by 3-5 points
Comparison of pain relief according Whatkins scale | 24 months
  Improvement on the Whatkins scale by 1-2 points

CONTACTS AND LOCATIONS:
Overall Officials: Aslan Valiev, PhD, Principal Investigator — N.N. Blokhin NMRCO; Pavel Kononets, PhD, Principal Investigator — N.N. Blokhin NMRCO
Locations (1):
- Federal State Budgetary Institution "N.N. Blokhin National Medical Research Center of Oncology" оf the Ministry of Health of the Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: official site — https://www.ronc.ru/about/struktura/niiko/ooo/hn1/
- See also: russian surcoma group site — https://sarcomarus.ru/